CLINICAL TRIAL: NCT02123355
Title: The Effect of Dexmedetomidine to Cognition of Geriatrics in Prolonged Surgery,A Randomized Controlled Study
Brief Title: The Effect of Dexmedetomidine to Cognition of Geriatrics in Prolonged Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaanxi Provincial People's Hospital (Other)
Collaborators: Chinese Medical Association (Network)
Responsible Party: Principal Investigator, Yang Li, Anesthesiologist, Shaanxi Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPPHA01
Record Dates: First submitted 2014-04-20; First posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Cognitive Ability, General; Brain Injury
MeSH Terms: conditions — Brain Injuries | interventions — Intubation; Sevoflurane; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine is given at 0.5μg/kg/h by continuous infusion and is stopped to given 30 minutes before the surgery is over.
  Interventions: Drug: Induction of anesthesia; Procedure: Intubation; Drug: Sevoflurane, remifentanil ,vecuronium; Drug: Dexmedetomidine
- Normal saline (Sham Comparator): Normal saline is given at 0.5μg/kg/h by continuous infusion and is stopped to given 30 minutes before the surgery is over.
  Interventions: Drug: Induction of anesthesia; Procedure: Intubation; Drug: Sevoflurane, remifentanil ,vecuronium; Drug: Placebo

INTERVENTIONS:
Drug: Induction of anesthesia — Midazolam 0.05 mg/kg、Propofol 1.0 mg/kg、Sufentanyl 3μg/kg、Victracurium 0.1 mg/kg sequential intravenous injection
Procedure: Intubation — After muscle relaxed and loss of eyelash reflex of the patients, intubation is done,then mechanical ventilation is performed, and maintain the PETCO2于35~40 mmHg，pulse oxygen saturation is more than 95%.
Drug: Sevoflurane, remifentanil ,vecuronium — Sevoflurane（1%-2%）is inspirated, and remifentanil 0.1-0.5μg/kg//min is continuously pumped,vecuronium 0.03 mg/kg is injected intermittently.
Drug: Dexmedetomidine — Dexmedetomidine is given at 0.5μg/kg/h by continuous infusion and is stopped to given 30 minutes before the surgery is over.
  Arms: Dexmedetomidine
Drug: Placebo — Normal saline is given at 0.5μg/kg/h by continuous infusion and is stopped to given 30 minutes before the surgery is over.
  Arms: Normal saline

SUMMARY:
The incidence of postoperative cognitive dysfunction (POCD) is high and POCD affect the life quality and the prognosis of patients. Geriatrics is the independent risk factor of POCD, and POCD is also correlated with many other factors such as type of surgery, the duration of anesthesia and the anesthesia drugs used et al. So, the prevention and treatment of POCD in geriatrics is important.

Dexmedetomidine is found to have the effect of neuro-protection, but it is controversy whether Dexmedetomidine has the effect of neuro-protection in geriatrics, especially the prolonged surgery.

The purpose of this study is to explore the effect of Dexmedetomidine to the cognitive function at prolonged surgery in geriatrics in geriatrics.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Scheduled for elective abdominal surgery
3. Age≥65 yrs
4. Weight is within the range of ±20% of standard weight [standard weight=Height(cm)-80)×70﹪ for male and(Height(cm)-70)×60﹪] for female
5. American society of anesthesia classification I~III
6. Expected time of surgery is more than 4 hours -

Exclusion Criteria:

1. Systolic blood pressure≥180 mm Hg or <90 mm Hg，diastolic blood pressure≥110 mm Hg or < 60 mm Hg；
2. Serious cardiac,liver,kidney,lung, endocrine disease or sepsis.
3. Allergy to trial drug or other contraindication；
4. Difficult airway occurred before,or difficult airway possibly occurred and difficult to extubation
5. History of mental illness and cerebral vascular disease
6. History of unstable angina or myocardial infarction
7. Education level<7 yrs
8. Factors existed that affect cognition assessment such as language, visual sense,auditory sense disorders.
9. Abuse of narcotic analgesia or suspected;
10. Neuromuscular diseases;
11. Mentally unstable or has a mental illness;
12. Pregnant or breast-feeding women;
13. Attended other trial past 30 days; -

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in cognitive function at 7 days | Baseline, the 7th day after the surgery
  1. Modified Newman scale to assess the cognitive function, including five tests.
  2. The quiet environment, enough daylight, no disturb is needed when the modified Newman scale is done. All the five tests are finished within 30 min.
  3. all the score of each test of all the patients assessed before the surgery is calculated, then get the standard variation, the score of each subject of each test is compared with the standard deviation, if one or more stand deviation decrease, then the cognitive function is considered as deterioration .
  4. When 2 or more of the tests is considered as deterioration, then the patients is diagnosed as Post Operation Cognitive Dysfunction (POCD).

SECONDARY OUTCOMES:
Brain injury assessment | From entering the operating room to 48 hours after the surgery
  1. 2 ml blood sample is collected at 8 time points including before surgery,the right moment,2 hr and 4 hr after the induction, the right moment,12,24 and 48 hours after the surgery.
  2. The serum level of C-reaction protein(CRP),tumor necrosis factor(TNF-α)、interleukin-6（IL-6）,interleukin-10（IL-10) is tested using immunohistochemical double antibody sandwich enzyme-linked immunosorbent assay (ELISA)
Inflammatory responsive assessment | From entering the operating room to 48 hours after the surgery
  1. 2 ml blood sample is collected at 8 time points including before surgery,the right moment,2 hr and 4 hr after the induction, the right moment,12,24 and 48 hours after the surgery.
  2. The concentration of protein S100B（S100B）and neuron specific enolase (NSE）in serum is tested using immunohistochemical double antibody sandwich enzyme-linked immunosorbent assay (ELISA).
Heart rate | From the induction of anesthesia to the right moment of extubation, up to 1 day.
  Heart rate are monitored every 15 min from the induction of anesthesia to the right moment of extubation.
Depth of anesthesia | From the induction of anesthesia to the right moment of extubation, up to 1 day.
  Bispectral index(BIS) monitor are performed every 15 min from the induction of anesthesia to the right moment of extubation.
Recovery of anesthesia | From the induction of anesthesia to the right moment of extubation, up to 1 day.
  Time of anesthetic ceased,time of call to open eyes,time to extubation, time to leave the PACU are recorded.
Central venous pressure(CVP) | From the induction of anesthesia to the right moment of extubation, up to 1 day.
  Central venous pressure(CVP) are monitored every 15 min from the induction of anesthesia to the right moment of extubation.
Blood pressure | From the induction of anesthesia to the right moment of extubation, up to 1 day.
  systolic blood pressure, Diastolic blood pressure are monitored every 15 min from the induction of anesthesia to the right moment of extubation.
Respiration rate | From the induction of anesthesia to the right moment of extubation, up to 1 day.
  Respiration rate are monitored every 15 min from the induction of anesthesia to the right moment of extubation.
Pulse blood oxygen saturation | From the induction of anesthesia to the right moment of extubation, up to 1 day.
  Pulse blood oxygen saturation are monitored every 15 min from the induction of anesthesia to the right moment of extubation.
Number of Participants with Serious and Non-Serious Adverse Events | Up to 7 days